CLINICAL TRIAL: NCT05199389
Title: Evaluating the Efficacy of Photobiomodulation Therapy in the Management of Chemotherapy-induced Peripheral Neuropathy: a Pilot Trial
Brief Title: Photobiomodulation Therapy in the Prevention and Management of Chemotherapy-Induced Peripheral Neuropathy
Acronym: NeuroLight
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/155
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Photobiomodulation therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PBM1 group (Experimental): The patients allocated to the first PBM-group will receive six PBM sessions of 6 J/cm² over three weeks (2x/week).
  Interventions: Device: Multiwave Locked System® (M6 laser, ASA srl, Arcugnano (VI), Italy)
- PBM2 group (Experimental): The patients allocated to the first PBM-group will receive six PBM sessions of 8 J/cm² over three weeks (2x/week).
  Interventions: Device: Multiwave Locked System® (M6 laser, ASA srl, Arcugnano (VI), Italy)

INTERVENTIONS:
Device: Multiwave Locked System® (M6 laser, ASA srl, Arcugnano (VI), Italy) — MLS® Laser M6 is a PBM device that allows the patients to be treated in various positions, either sitting, lying down or at a distance, without risk of contamination. Treatment times are carefully calibrated to deliver the best possible energy dose to the tissue being treated.

SUMMARY:
This study aims to investigate the effectiveness of photobiomodulation therapy (PBM) in the management of chemotherapy-induced peripheral neuropathy (CIPN). Therefore, the hypothesis is that PBM can reduce the severity of CIPN in cancer patients, increasing the patient's quality of life.

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) is one of the common complications of cancer treatment and involves paresthesia, numbness and/or burning pain in distal limbs. This condition has a high health impact because it is associated with psychological distress, fall risk, and poor sleep quality. Furthermore, it impairs patients' daily activities and thereby decreases their quality of life. The overall incidence of CIPN is approximately 68% in the first month after chemotherapy. The available evidence for preventive and therapeutic options for CIPN is limited. Therefore, only symptom management based on pharmacological and/or physical therapy is applied with limited success. Our research group showed that photobiomodulation (PBM) has the potential to reduce the development of CIPN in breast cancer patients (unpublished data). PBM uses visible and/or (near)-infrared light at a low power produced by laser diodes or light-emitting diodes (LED) to stimulate tissue repair and reduce inflammation and (neuropathic) pain. The aim of this project is to evaluate the effectiveness of PBM in the management of CIPN in general.

ELIGIBILITY:
Inclusion Criteria:

* Finished one of the following types of chemotherapy: paclitaxel, docetaxel, oxaliplatin, cisplatin, vincristine, thalidomide and/or bortezomib.
* Diagnosed with CIPN
* Age 18 years or above
* Have no documented or observable psychiatric or neurological disorders that might interfere with study participation (e.g., dementia or psychosis)
* Dutch-speaking
* Signed informed consent

Exclusion Criteria:

* Taking stable doses of medication on prescription for peripheral neuropathy. Related medications are: gabapentin, pregabalin (Lyrica), nortriptyline, amitriptyline, duloxetine (Cymbalta), and venlafaxine.
* Severe or unstable cardio- respiratory or musculoskeletal disease
* Interruption of more than two consecutive laser treatments
* Dark brown or black skin pigmentation (described as skin type VI in the Fitzpatrick scale)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2028-11-10 (Estimated)

PRIMARY OUTCOMES:
Modified total neuropathy score (mTNS) | Baseline
  The mTNS is a clinically applicable, sensitive screening tool for CIPN. The score ranges from 0 to 24, with a higher score indicating a higher level of neuropathy.
Modified total neuropathy score (mTNS) | End of PBM (three weeks post-baseline)
  The mTNS is a clinically applicable, sensitive screening tool for CIPn. The score ranges from 0 to 24, with a higher score indicating a higher level of neuropathy.
Modified total neuropathy score (mTNS) | Three weeks post-PBM
  The mTNS is a clinically applicable, sensitive screening tool for CIPN. The score ranges from 0 to 24, with a higher score indicating a higher level of neuropathy.
Pain score | Baseline
  The patients' pain due to CIPN will be evaluated by using a numerical rating scale (NRS). The score ranges from 0 to 10, with a higher score indicating a higher level of pain.
Pain score | End of PBM (three weeks post-baseline)
  The patients' pain due to CIPN will be evaluated by using a numerical rating scale (NRS). The score ranges from 0 to 10, with a higher score indicating a higher level of pain.
Pain score | Three weeks post-PBM
  The patients' pain due to CIPN will be evaluated by using a numerical rating scale (NRS). The score ranges from 0 to 10, with a higher score indicating a higher level of pain.
Mobility score | Baseline
  The mobility of the patients will be measured using the six minute walk test. This test measures the distance the patient can walk in six minutes and compares it to the normal value for their age and BMI.
Mobility score | End of PBM (three weeks post-baseline)
  The mobility of the patients will be measured using the six minute walk test. This test measures the distance the patient can walk in six minutes and compares it to the normal value for their age and BMI.
Mobility score | Three weeks post-PBM
  The mobility of the patients will be measured using the six minute walk test. This test measures the distance the patient can walk in six minutes and compares it to the normal value for their age and BMI.

SECONDARY OUTCOMES:
Quality of life score | Baseline
  The Functional Assessment of Cancer Therapy/ Gynecologic Oncology Group Neurotoxicity (FACT/GOG-NTX) is a validated patient questionnaire to test the quality of life of the patients with CIPN. The score ranges from 0 to 152, with a higher score indicating a lower quality of life.
Quality of life score | End of PBM (three weeks post-baseline)
  The Functional Assessment of Cancer Therapy/ Gynecologic Oncology Group Neurotoxicity (FACT/GOG-NTX) is a validated patient questionnaire to test the quality of life of the patients with CIPN. The score ranges from 0 to 152, with a higher score indicating a lower quality of life.
Quality of life score | Three weeks post-PBM
  The Functional Assessment of Cancer Therapy/ Gynecologic Oncology Group Neurotoxicity (FACT/GOG-NTX) is a validated patient questionnaire to test the quality of life of the patients with CIPN. The score ranges from 0 to 152, with a higher score indicating a lower quality of life.
Satisfaction score | Baseline
  The patients' global satisfaction with the PBM therapy will be evaluated using a NRS from 0 (minimum score) to 10 (maximum score).
Satisfaction score | End of PBM (three weeks post-baseline)
  The patients' global satisfaction with the PBM therapy will be evaluated using a NRS from 0 (minimum score) to 10 (maximum score).
Satisfaction score | Three weeks post-PBM
  The patients' global satisfaction with the PBM therapy will be evaluated using a NRS from 0 (minimum score) to 10 (maximum score).

OTHER OUTCOMES:
General patient-, disease-, and treatment-related information | Baseline
  General and medical information will be collected through a short patient questionnaire in order to assess intrinsic risk factors (e.g. age and smoking history). Information regarding the disease- and treatment-related risk factors will be collected through medical records (e.g., tumour type and stage).
General patient-, disease-, and treatment-related information | End of PBM (three weeks post-baseline)
  General and medical information will be collected through a short patient questionnaire in order to assess intrinsic risk factors (e.g. age and smoking history). Information regarding the disease- and treatment-related risk factors will be collected through medical records (e.g., tumour type and stage).
General patient-, disease-, and treatment-related information | Three weeks post-PBM
  General and medical information will be collected through a short patient questionnaire in order to assess intrinsic risk factors (e.g. age and smoking history). Information regarding the disease- and treatment-related risk factors will be collected through medical records (e.g., tumour type and stage).
Cancer relapse or recurrence | One year post chemotherapy
  The possibility of cancer relapse or recurrence will be evaluated using the patients' medical records.
Cancer relapse or recurrence | Two years post chemotherapy
  The possibility of cancer relapse or recurrence will be evaluated using the patients' medical records.
Cancer relapse or recurrence | Three years post chemotherapy
  The possibility of cancer relapse or recurrence will be evaluated using the patients' medical records.
Cancer relapse or recurrence | Four years post chemotherapy
  The possibility of cancer relapse or recurrence will be evaluated using the patients' medical records.
Cancer relapse or recurrence | Five years post chemotherapy
  The possibility of cancer relapse or recurrence will be evaluated using the patients' medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Mebis, Prof. Dr., Principal Investigator — Jessa Hospital
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium